CLINICAL TRIAL: NCT00304655
Title: Multicenter, Single Group Study of Aripiprazole Efficacy and Safety in the Acute Psychosis Treatment of Schizophrenia, Schizophreniform Disorder and Schizoaffective Disorder.
Brief Title: Acute Psychosis Treatment in the Long Term, Unitary Group Study (APLUS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Korea Otsuka Pharmaceutical Co.,Ltd., Korea Otsuka Pharmaceutical Co.,Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOP-010401
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective disorder; Aripiprazole
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The purpose of this study is to prove safety and efficacy of aripiprazole.

DETAILED DESCRIPTION:
This study was designed to prove safety and efficacy of aripiprazole in the treatment of acutely relapsed patients with diagnoses of schizophrenia or schizoaffective disorder in Korea and to confirm the maintenance of efficacy and safety during maintenance period and the changes in emotional factors and social functions.

After administering 15 mg/day of aripiprazole for two weeks, the test may change the dose within the range of 10 mg and 30 mg per day by clinical judgment. (Medication duration: 8 weeks (acute phase) + 18 weeks (maintenance phase)] + 26 weeks (extension phase), *total 52 weeks)

ELIGIBILITY:
Inclusion Criteria:

1. Schizophrenia or schizoaffective disorder patients as defined by the DSM-IV criteria having an acute relapse
2. 18 to 65 years
3. Males and females (females of child bearing potential must use acceptable contraception and must not be pregnant and lactating; females of child-bearing potential must have negative serum pregnancy test)
4. Randomization to this study must occur no more than four weeks following the day of initiation of treatment for the present episode/relapse.
5. Should have a total PANSS score of at least 60. In addition, patients should have scores of at least 4 ("moderate") on any two of the four PANSS items that constitute the psychotic item subscale (hallucinatory behavior, delusions, conceptual disorganization, and suspiciousness).
6. Patients must be able to be rated reliably on the battery of psychiatric and movement rating scales required by the protocol.
7. Patients eligible to enter the study must sign an informed consent form.

Exclusion Criteria:

1. Patients who are violent
2. Patients who, in the opinion of the investigator, have serious suicidal ideation
3. Patients who are liable to serious suicide attempt, by clinical judgment
4. Patients who currently have a psychiatric diagnosis other than schizophrenia, schizophrenic form disorder or schizoaffective disorder requiring pharmacotherapy
5. Patients who have any of the following neurologic diagnoses: migraine, epilepsy, Parkinson's disease, Alzheimer's disease, multiple sclerosis, residual of stroke, transient cerebral ischemic attacks, "cerebral palsy" or any other condition that requires intermittent or maintenance treatment, or which is manifested by any abnormality on neurologic examination
6. Patients who must continue to take, or who may potentially need to take, during this study, any of the following concomitant medication, which could cause unwanted drug-to-drug interactions or which could confound the analysis of antipsychotic effectiveness: Tegretol (carbamazepine), Depakene Depakote (valproic acid or sodium valproate or divalproate sodium), Lithium carbonate and lithium citrate
7. Patients under treatment of schizophrenia : those who had taken antipsychotic drugs (consta) before randomization
8. Patients who must continue to take, during this study, drugs or substances known as strong suppressive agents of microsomal enzyme CYP2D6
9. Patients with any gastrointestinal resection, stomach stapling, or any other condition that may impair the absorption of the study medication
10. Patients who currently meet the DSM-IV criteria for psychoactive substance dependence or patients with a history of substance or alcohol dependence (according to the DSM-IV criteria) within one month prior to the beginning of the study
11. Patients having any somatic condition whose symptoms or physical signs could be misinterpreted as signs or symptoms of psychosis or as adverse effects from antipsychotic medications.
12. Patients with any acute or unstable medical condition requiring pharmacotherapy
13. Patients with any abnormal laboratory test result as judged by investigator
14. Patients who have participated in any previous aripiprazole clinical study
15. Patients having taken an investigational drug within the four weeks which precede the start of placebo washout

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-07; Primary Completion 2006-05 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
PANSS-total score (at screening, week 1, 2, 3, 4, 6, 8, 12, 16, 26, 40, 52)

SECONDARY OUTCOMES:
[Efficacy] PANSS-positive, PANSS-negative, CGI-severity score (at screening, week 1, 2, 3, 4, 6, 8, 12, 16, 26, 40, 52)
[Safety] AEs (at baseline, week 1, 2, 3, 4, 6, 8, 12, 16, 26, 40, 52)
SAS, AIMS, Barnes (at baseline, week 1, 2, 3, 4, 6, 8, 12, 16, 26, 40, 52)
vital signs (at screening, baseline, week 1, 2, 3, 4, 6, 8, 12, 16, 26, 40, 52)
body weight (at screening, baseline, week 1, 2, 3, 4, 6, 8, 12, 16, 26, 40, 52)
electrocardiogram (ECG) (at screening & week 8)
serum prolactin concentration (at screening & week 8)
routine laboratory test (at screening & week 8)
urinalysis (at screening & week 8)
Pharmacokinetic is evaluated by concentration of aripiprazole in blood (at Week 3, 4, 6, 8).

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Su Kwon, Prof., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea